CLINICAL TRIAL: NCT06286150
Title: Efficacy and Safety of Single-port Surgical Robot System in Thoraic Surgery: A Prospective, Single Center Study
Brief Title: Efficacy and Safety of Single-port Surgical Robot System in Thoraic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Director, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-2023-087(QX)-03
Record Dates: First submitted 2024-02-15; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
Keywords: surgical robot system; efficacy; safety; thoracic surgery
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-port robot group (Experimental)
  Interventions: Procedure: Surgical robot system

INTERVENTIONS:
Procedure: Surgical robot system — SHURUI Single-port surgical robot system

SUMMARY:
Robotic surgical systems have become a promising surgical assistance system, with unique advantages such as 3D high-definition visual system, highly flexible wrist-jointed instruments, and automatic fitering of hand tremors. Robotic surgical systems is applied in various fields including urology, general surgery, cardiothoracic surgery, head and neck surgery, and gynecology. Currently, the Da Vinci surgical robot system is the most widely used robot system globally. However, the Da Vinci robot system for single-port laparoscopic surgery has not yet been launched in China. Therefore, the investigators conduct a prespective, single-center study to evaluate the efficacy and safety of single-port surgical robot system in thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years, regardless of gender.
* Patients who require endoscopic surgical treatment and have indications for lung segment/lobe resection; for pre-trial subjects, there is no restriction on the type of procedure, and inclusion is based on the investigator's judgment of having indications for thoracic surgery.
* Preoperative ASA classification of I-III.
* Voluntary participation in the clinical trial and willingness to provide informed.

consent, either by the subject or their guardian.

* Willingness to cooperate and complete trial follow-up and related examinations.

Exclusion Criteria:

* Patients with a history of thoracic surgery or previous history of other malignant tumors deemed unsuitable for inclusion by the investigator.
* Patients with severe comorbidities (cardiac, pulmonary, hepatic, cerebral, renal diseases) or physical weakness who cannot tolerate general anesthesia or surgery.
* Patients with severe bleeding tendencies or coagulation disorders.
* Patients in the active phase of infectious diseases or with other severe non-communicable infections.
* Patients positive for Human Immunodeficiency Virus (HIV) antibodies or syphilis seropositive patients.
* Patients with a suspected or confirmed alcohol, drug, or substance addiction.
* Patients with a history of epilepsy, mental illness, or cognitive impairment.
* Women who are pregnant, breastfeeding, or planning to become pregnant during the trial period.
* Participation in other interventional clinical trials within 3 months prior to signing the informed consent form.
* Other situations in which the investigator deems inappropriate for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative conversion rate | Within 1 day after surgery
  The conversion from a single-port laparoscopic surgery system to other surgical Instrument control systems, such as traditional thoracoscopy or open surgery.
Surgical complications rate | 30 days after surgery
  The incidence rate of instrument-related or potentially instrument-related surgical complications meeting Clavien-Dindo grade 3 or above criteria from the time of incision

SECONDARY OUTCOMES:
Intraoperating bleeding volume | Within 1 day after surgery
  The amount of intraoperative bleeding from the start to the end of the surgery in the study subjects
Surgical time | Within 1 day after surgery
Length of hospital admissions | Within 30 day after surgery
  The total number of days of hospitalization from the day of surgery to discharge for the study subjects.
  If a subject is admitted in the afternoon or discharged in the morning, the day of admission or discharge is recorded as 0.5 days.
Postoperative wound pain score | 1, 24 and 72 hours after surgery
  Assessment will be conducted using the Numerical Rating Scale (NRS)
Surgeon satisfaction | Within 4 hours after surgery
  The surgeon satisfaction survey questionnaire consists of two parts: performance-related (12 questions) and surgeon comfort-related ratings (8 questions). The scoring criteria are as follows: Each question is scored on a scale of 1-5, with a maximum score of 5. The total score is out of 100
Adverse events | Within 1 day after surgery
  Incidence of adverse events (AE), serious adverse events (SAE), and overall surgical complication rate (evaluated using the Clavien-Dindo grading system)
Rate of re-admission to hospital | 30 days after discharge
Rate of reoperation | 30 days after surgery
Postoperative mortality | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China